CLINICAL TRIAL: NCT05457283
Title: An 18-month, Open-label, Single-arm Safety Extension Study of an age-and Bodyweight-adjusted Oral Finerenone Regimen, in Addition to an ACEI or ARB, for the Treatment of Children and Young Adults From 1 to 18 Years of Age With Chronic Kidney Disease and Proteinuria
Brief Title: A Study to Learn More About How Safe the Study Treatment Finerenone is in Long-term Use When Taken With an ACE Inhibitor or Angiotensin Receptor Blocker Over 18 Months of Use in Children and Young Adults From 1 to 18 Years of Age With Chronic Kidney Disease and Proteinuria
Acronym: FIONA OLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20186; 2023-504885-50-00 (Registry Identifier: CTIS (EU)); 2021-002905-89 (EudraCT Number)
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Proteinuria; Children
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Finerenone Open-Label safety Extension (Experimental): Participants will receive finerenone treatment.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Finerenone in different doses, treatment duration will be 540 ±7 days.

SUMMARY:
Researchers are looking for a better way to treat children who have chronic kidney disease (CKD), which is long-term kidney disease, and proteinuria, a condition in which a person´s kidneys leak protein into the urine.

The kidneys filter waste and fluid from the blood to form urine. In children with CKD, the kidney´s filters do not work as well as they should. This can lead to accumulation of waste and fluid in the body and proteinuria. CKD can lead to other medical problems, such as high blood pressure, also known as hypertension. Vice versa, hypertension and proteinuria can also contribute to worsening of CKD. Therefore, the treatment of CKD aims to control blood pressure and proteinuria. There are treatments available for doctors to prescribe to children with CKD and hypertension and/or proteinuria. These include "angiotensin-converting enzyme inhibitors" (ACEI) and "angiotensin receptor blockers" (ARB). Both ACEI and ARB can help improve kidney function by reducing the activity of the renin-angiotensin-aldosterone system (RAAS). The RAAS is a system that works with the kidneys to control blood pressure and the balance of fluid and electrolytes in the blood. In people with CKD, the RAAS is often too active, which can impair the ability of the kidneys to work properly and cause hypertension and proteinuria. However, ACEI or ARB treatment alone does not work for all patients with CKD as they only target the angiotensin part of the renin-angiotensin-aldosterone system.

The study treatment, finerenone, is expected to help control RAAS overactivation together with an ACEI or ARB.

So, the researchers in this study want to learn more about whether finerenone given in addition to either an ACEI or ARB can help their kidney function.

The main purpose of this study is to learn how safe the treatment is when used of finerenone in addition to an ACEI or ARB in long-term.

To see how safe the treatment is, the study team will collect information on medical problems which are also known as "treatment emergent adverse events" (TEAEs). And they will also collect levels of an electrolyte called potassium in the blood by taking blood samples, and measure blood pressure during the study.

The secondary purpose of this study is to learn how well long-term use of finerenone can reduce the amount of protein in the participants' urine and benefit kidney function when taken with standard of care.

To see how the treatment works, the study team will collect participants' urine samples to assess urinary albumin-to-creatinine ratio (UACR) and urinary protein-to-creatinine ratio (UPCR), which are important assessments for calculating the level of protein in the urine. Researchers will also collect blood samples to analyze serum creatinine and calculate estimated glomerular filtration rate (eGFR). A significant decline in eGFR indicates worsening kidney function.

The study will include participants who had previously participated in FIONA study (NCT05196035). The participants will be aged from 1 year up to 18 years.

The participants will be in the study for approximately 19 months. They will take study treatment for up to 18 months and will be follow up for 1 month. During this period, at least 12 visits are planned for patients who newly start finerenone, and at least 8 visits for patients who already received finerenone.

In the visit, the study team will:

* have their blood pressure, heart rate, temperature, height and weight measured
* have blood and urine samples taken
* have physical examinations
* have their heart examined by an electrocardiogram and echocardiography (a sonogram of the heart)
* answer questions about their medication and whether they have any adverse events, or have their parents or guardian's answer
* answer questions about how they are feeling, or have their parents or guardian's answer
* answer question about how they like the study medication, or have their parents or guardian's answer The doctors will keep track of any adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

The doctors will check the participants' health about 30 days after the participants take their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥1 year to 18 years of age, at the time of signing the informed consent/assent.
* Prior participation in the finerenone Phase 3 study FIONA (19920) and not permanently discontinued from treatment by the end of treatment (EoT) visit in FIONA.
* Participants must have a clinical diagnosis of chronic kidney disease (CKD) at Visit 1 which is defined as

  * CKD stages 1-3 (estimated glomerular filtration rate [eGFR] ≥30 mL/min/1.73m^2) for children ≥1 year to <19 years of age at FIONA EoT and at Visit 1
* Treated with an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) at optimized doses defined as maximally tolerable doses within the recommended dose range according to guidelines on blood pressure (BP) management, unchanged for at least 30 days prior to Visit 1.
* K+ ≤5.0 mmol/L for children ≥2 years of age at both FIONA EoT and Visit 1, and ≤5.3 mmol/L for children <2 years of age at both FIONA EoT and Visit 1
* Participants who have reached legal age of consent: Capable of giving signed informed consent.
* Participant is able to receive enteral feeding (solid food, bottle or cup fed, feeding through nasogastric or gastric feeding tubes) with or without breastfeeding.

Exclusion Criteria:

* Planned urological surgery expected to influence renal function
* Patients who are candidates for renal transplantation, i.e., a kidney transplantation scheduled within the study time frame
* Systemic hypertension Stage 2 defined according to institutional guidelines on BP management at Visit 1.
* Systemic hypotension defined as symptomatic hypotension or a mean systolic BP below the 5th percentile for age, sex and height but no lower than 80 mmHg for participants <18 years and symptomatic hypotension or a mean systolic blood pressure (SBP) <90 mmHg in participants ≥18 years at Visit 1.
* Known hypersensitivity to the study treatment (active substance or excipients)
* Severe hepatic insufficiency defined by e.g. Child-Pugh C or analogous scores.
* Participants using rituximab, cyclophosphamide, abatacept, or intravenous glucocorticoids
* Concomitant therapy with a mineralocorticoid receptor antagonist (MRA)(eplerenone, spironolactone, esaxerenone, canrenone), any renin inhibitor (aliskiren, enalkiren, remikiren), any sodium-glucose co-transporter-2 (SGLT2) inhibitor (SGLT2i), sacubitril/valsartan combination (ARNI), or potassium-sparing diuretic (amiloride, triamterene)
* Concomitant therapy with both ACEI and ARBs together
* Concomitant therapy with strong cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors, moderate or strong CYP3A4 inducers
* Previous assignment to treatment during this study
* Simultaneous participation in another interventional clinical study (e.g., Phase 1 to 4 clinical studies).
* Any suspected (serious) adverse event related to study intervention which led to permanent discontinuation during the FIONA study.
* Pregnant or breastfeeding or intention to become pregnant during the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2029-01-28 (Estimated); Study Completion 2029-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse event (TEAEs) | Up to 550 days
Change in serum potassium levels from baseline to Day 540±7 | Up to 547 days
Change in systolic blood pressure (SBP) from baseline to Day 540±7 | Up to 547 days

SECONDARY OUTCOMES:
Change in urinary protein-to-creatinine ratio (UPCR) from baseline to Day 540±7 | Up to 547 days
Change in urinary albumin-to-creatinine ratio (UACR) from baseline to Day 540±7 | Up to 547 days
Change in estimated glomerular filtration rate (eGFR) from baseline to Day 540±7 | Up to 547 days

CONTACTS AND LOCATIONS:
Locations (177):
- United States (18):
  - Phoenix Children's Hospital | Main - Transplant Department, Phoenix, Arizona
  - Cedars-Sinai Samuel Oschin Cancer Center, Los Angeles, California
  - Lucille Packard Children's Hospital Stanford - Pediatric Nephrology, Palo Alto, California
  - Rady Children's Hospital San Diego - Cardiology, San Diego, California
  - Children's National Hospital - Nephrology, Washington D.C., District of Columbia
  - Memorial Transplant Institute - Pediatric Nephrology, Hollywood, Florida
  - Emory University Hospital/Children's Healthcare of Atlanta - Nephrology, Atlanta, Georgia
  - University of Iowa Health Care Medical Center - Nephrology, Iowa City, Iowa
  - The Charlotte R. Bloomberg Children's Center Building - Nephrology, Baltimore, Maryland
  - Boston Children's Hospital - Main Campus - Nephrology, Boston, Massachusetts
  - Children's Mercy Hospital Kansas City - Nephrology, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center | Division of Nephrology and Hypertension, Cincinnati, Ohio
  - Cleveland Clinic | Pediatric Nephrology, Cleveland, Ohio
  - OHSU Doernbecher Children's Hospital - Neurology, Portland, Oregon
  - Children's Hospital of Philadelphia - Nephrology, Philadelphia, Pennsylvania
  - University Hospital - San Antonio - Pediatric Nephrology, San Antonio, Texas
  - Eccles Primary Children's Outpatient Services - Nephrology, Salt Lake City, Utah
  - Seattle Children's Hospital - Nephrology, Seattle, Washington
- Argentina (8):
  - Hospital de Niños Sor María Ludovica, La Plata, Buenos Aires
  - Hospital General de Ninos Ricardo Gutierrez | Pediatric Nephrology Department, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Centro de Rehabilitacion Cardiovascular | San Luis, Argentina, San Luis, San Luis Province
  - Clinica de Nefrologia, Urologia y Enfermedades Cardiovascualares | Santa Fe, Argentina, Santa Fe, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Pediatría Juan P. Garrahan, Buenos Aires
  - Hospital General de Ninos Pedro de Elizalde | Nephrology Department, Ciudad Autonoma de Buenos Aire
  - Many Locations, Multiple Locations
- Australia (3):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital Melbourne, Parkville, Victoria
- Austria (5):
  - Medizinische Universität Graz, Graz, Styria
  - Kepler Universitätsklinikum Campus IV, Innsbruck, Tyrol
  - Uniklinikum Salzburg - Landeskrankenhaus, Vienna, Vienna
  - Universitätsklinikum AKH Wien, Vienna, Vienna
  - Many Locations, Multiple Locations
- Belgium (6):
  - Huderf / Ukzkf, Bruxelles - Brussel
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Gasthuisberg - Pediatric Nephrology, Leuven
  - CHC Montlégia - Pediatrics, Liège
  - Many Locations, Multiple Locations
- Brazil (6):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Pequeno Principe, Curitiba, Paraná
  - Hosp Clínicas Facult. Med. de Ribeirão Preto / USP, Ribeirão Preto/SP, São Paulo
  - Hospital Infantil Sabará - Instituto PENSI - Pesquisa e Ensino em Saúde Infantil, São Paulo, São Paulo
  - Hospital PUC-Campinas | Centro de Pesquisa Clínica Sao Lucas, São Paulo, São Paulo
  - Instituto da Crianca e do Adolescente, São Paulo
- Bulgaria (3):
  - UMHAT Sveti Georgi, Plovdiv
  - SHATPD "Prof. Ivan Mitev", Sofia
  - MHAT prof. Stoyan Kirkovitch AD, Stara Zagora
- Canada (3):
  - Alberta Children's Hospital - Nephrology Clinic, Calgary, Alberta
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Czechia (3):
  - Many Locations, Multiple Locations
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Fakultní nemocnice Motol a Homolka, Pracovište MOTOL, Prague
- Denmark (4):
  - Aarhus Universitetshospital - Børn og Unge, Århus N
  - Rigshospitalet - Børn og Unge, Copenhagen
  - Many Locations, Multiple Locations
  - Odense Universitetshospital - HC Andersen Børne og Ungehospital, Odense C
- Finland (4):
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Uusi lastensairaala, nefrologia, Helsinki
  - Many Locations, Multiple Locations
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS) - Lasten lääketutkimuskeskus PeeTU, Tampere
  - Turun yliopistollinen keskussairaala, Turku
- France (7):
  - CHU bordeaux - Hopital Pellegrin, Bordeaux
  - CHU de Lyon - Hopital Femme Mère Enfant, Bron
  - Hopital Arnaud de Villeneuve CHU Montpellier, Montpellier
  - Many Locations, Multiple Locations
  - Hopital Robert Debre, Paris
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg
  - Hôpital des Enfants, Toulouse
- Germany (9):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Medizinische Hochschule Hannover (MHH) | Zentrum Innere Medizin | Klinik fuer Kardiologie und Angiologie, Hanover, Lower Saxony
  - Kindernierenzentrum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Charité / Pädiatrie, Berlin
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
  - Many Locations, Multiple Locations
- Greece (6):
  - Children's Hospital of Athens P&A Kyriakou - Pediatric Nephrology Department, Athens
  - Children's Hospital of Athens Agia Sofia - Pediatric Nephrology Department, Athens
  - University General Hospital of Heraklion - Department of Paediatrics, Heraklion
  - University General Hospital Of Ioannina-Child Health Sector, Ioannina
  - Many Locations, Multiple Locations
  - Ippokratio General Hospital Of Thessaloniki-Pediatric Nephrology Unit, 3rd Department of Paediatrics, Thessaloniki
- Hungary (5):
  - Semmelweis University, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Many Locations, Multiple Locations
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- India (4):
  - Mavani Kidney Care, Ahmedabad
  - St. John's National Academy of Health Sciences, Bangalore
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, Delhi
  - NRS Medical college, Kolkata
- Israel (6):
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Wilf Children's Hospital Shaare Zedek Medical Center, Jerusalem
  - Many Locations, Multiple Locations
  - Health Corporation of Galilee Medical Center, Nahariya
  - Clalit Health Services Schneider Children's Medical Center, Petah Tikva
  - Dana-Dwek Children's Hospital, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Pediatria, Bologna, Emilia-Romagna
  - Ospedale Pediatrico Bambino Gesù - Nefrologia, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini - Nefrologia e Trapianto Rene, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Nefrologia e Dialisi Pediatrica, Trapianti di Rene, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Meyer IRCCS - Nefrologia e Dialisi, Florence
  - Many Locations, Multiple Locations
  - A.O.U. Città della Salute e della Scienza di Torino_Regina Margherita - Nefrologia Pediatrica, Torino
- Lithuania (4):
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Children's Hospital, Klaipėda
  - Many Locations, Multiple Locations
  - Vilnius University Hospital Santaros Klinikos Children's Hospital Paediatrics Centre, Vilnius
- Malaysia (5):
  - Hospital Tunku Azizah, Wilayah Persekutuan, Kuala Lumpur
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Hospital Selayang, Shah Alam, Selangor
  - Sunway Medical Centre, Subang Jaya, Selangor
  - Hospital Universiti Sains Malaysia, Kelantan
- Mexico (5):
  - Sitio Alfredo Chew Wong | Aguascalientes, Mexico, Aguascalientes, Agguascalientes
  - Hospital Infantil de México "Dr. Federico Gómez", México D.F., Mexico City
  - Instituto Nacional de Pediatría, México, D.F., Mexico City
  - Hospital Universitario "José Eleuterio González", Monterrey, Nuevo León
  - Instituto Veracruzano en Investigación Clinica SC, Veracruz
- Netherlands (3):
  - Universitair Medisch Centrum Groningen, Groningen
  - Many Locations, Multiple Locations
  - University Medical Center Utrecht, Utrecht
- Poland (7):
  - Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Many Locations, Multiple Locations
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego We Wroclawiu, Wroclaw
- Portugal (4):
  - Centro Clinico Academico Braga | Braga, Portugal, Braga
  - Hospital Pediátrico de Coimbra I ULS Coimbra, Coimbra
  - Hospital Santa Maria | Centro de Investigacao Clinica, Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
- South Korea (6):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang''yeogsi
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Many Locations, Multiple Locations
  - Korea University Guro Hospital, Seoul
- Spain (7):
  - Hospital Universitari Vall D Hebron | Nefrologia pediatrica, Barcelona
  - Hospital Sant Joan De Deu Barcelona | Nefrologia pediatrica, Barcelona
  - Hospital Universitario 12 De Octubre | Nefrologia pediatrica, Madrid
  - Hospital Universitario La Paz | Nefrologia pediatrica, Madrid
  - Hospital Universitario Regional De Malaga | Nefrologia pediatrica, Málaga
  - Many Locations, Multiple Locations
  - Hospital Universitario Virgen Del Rocio S.L. | Nefrologia pediatrica, Seville
- Sweden (4):
  - Skåne University Hospital, Lund
  - Many Locations, Multiple Locations
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Switzerland (4):
  - Universitäts-Kinderspital UKBB, Basel, Canton of Basel-City
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Hopital des Enfants HUG, Geneva
  - Many Locations, Multiple Locations
- Taiwan (6):
  - National Cheng Kung University Hospital, Tainan, TNN
  - Chang Gung Memorial Hospital (CGMH) - Kaohsiung Branch, Guishan
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (9):
  - Cukurova Univ. Tip. Fak. Balcali Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Baskent Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - T.C. Saglik Bakanligi Ankara Bilkent Sehir Hastanesi Noroloji ve Ortopedi Hastanesi Noroloji Bolumu, Ankara
  - Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatrics, Istanbul
  - Istanbul Universitesi Cerrahpasa - Cocuk Nefrolojisi, Istanbul
  - Marmara University Medical Faculty | Pediatric Nephrology, Istanbul
  - Many Locations, Multiple Locations
- United Kingdom (6):
  - Great Ormond Street Hospital for Children NHS Foundation Trust | Great Ormond Street Hospital - Clinical Research Facility, London, Greater London
  - Manchester University NHS Foundation Trust | Royal Manchester Children's Hospital - Clinical Research Facility, Manchester, Greater Manchester
  - Nottingham University Hospitals NHS Trust | Queens Medical Centre - Childrens Clinical Research Facility, Nottingham, Nottinghamshire
  - NHS Greater Glasgow and Clyde | Royal Hospital for Children - Glasgow Clinical Research Facility, Glasgow, Scotland
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - Many Locations, Multiple Locations

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.